CLINICAL TRIAL: NCT03123029
Title: Expanded Access to Venetoclax
Status: Available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C16-431; C19-920 (Other Grant/Funding Number: Abbvie); C20-485 (Other Grant/Funding Number: Abbvie)
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-04

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Multiple Myeloma; Acute Myeloid Leukemia (AML); Non-Hodgkin's Lymphoma; Acute Lymphoblastic Leukemia (ALL); Amyloidosis; Plasma Cell Leukemia
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Amyloidosis; Leukemia, Plasma Cell | interventions — venetoclax

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Venetoclax — Venetoclax will be administered orally.
  Other Names: ABT-199; GDC-0199

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to Venetoclax prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Exclusion Criteria:

* There are other suitable treatment options.
* The participant qualifies for ongoing clinical trials.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie